CLINICAL TRIAL: NCT00391677
Title: Effectiveness Trial of Attention Shaping for Schizophrenia
Brief Title: Attention Shaping Procedures for Improving Psychosocial Skills Among Adults With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH074650 (NIH); R01MH074650 (NIH); DATR A2-A1SZ
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: Cognitive Rehabilitation; Behavior Therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive social skills training with attention shaping procedures
  Interventions: Behavioral: Social skills training with attention shaping procedures
- 2 (Active Comparator): Participants will receive social skills training without attention shaping procedures
  Interventions: Behavioral: Social skills training without attention shaping

INTERVENTIONS:
Behavioral: Social skills training with attention shaping procedures — Social skills training with attention shaping procedures includes behavioral procedures to increase the frequency, intensity, and duration of attentive behaviors and to reduce the frequency of inattentive behaviors.
  Arms: 1
Behavioral: Social skills training without attention shaping — Social skills training without attention shaping is based on the UCLA Basic Conversation Skills Training Module, used without attention shaping procedures.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of attention shaping procedures in improving attentiveness and learning abilities in people undergoing psychosocial skills training treatment for schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a disabling mental disorder that can interfere with a person's ability to function both alone and in social situations. Various treatments have been effective in treating schizophrenia, including antipsychotic medications and cognitive therapy. Psychosocial skills training, a type of cognitive therapy, is often used to help people with schizophrenia cope with their condition and improve social functioning in day-to-day life. However, many individuals with schizophrenia experience difficulty paying attention, and this is a significant barrier to successful outcomes in psychosocial skills training interventions. Attention shaping procedures (ASP) is a behavioral intervention that helps individuals with impaired attention capacities to benefit from skills-based treatment. This study will evaluate the effectiveness of ASP in improving attentiveness and learning abilities in people undergoing psychosocial skills training treatment for schizophrenia.

Participants in this 5-month, single-blind study will be randomly assigned to ASP plus basic conversation skills training (BCS), which is a social skills training group, or BCS alone. Training sessions for both groups will be held when participants attend regular hospital visits. During the first month, participants will complete two sessions of interviews, self-report scales, and social and cognitive functional assessments. Over the next 3 months, training sessions for both groups will occur twice a week for approximately 1 hour. ASP sessions will focus on setting goals and increasing the quality and duration of participants' attentiveness during psychosocial interventions. BCS will train participants in the following five skill areas: recognizing verbal and non-verbal cues; starting a friendly conversation; keeping conversation going; ending a conversation politely; and incorporating all of these skills together. During the last month, participants will attend two interview sessions lasting approximately 4 hours each. One follow-up session will occur 6 months after completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, as confirmed by a diagnostic interview
* Has experienced difficulty paying attention while in groups during a treatment program, as determined by program staff
* Has experienced problems with social skills, as determined by program staff and study clinicians
* Social skill deficits, as determined by study clinicians

Exclusion Criteria:

* Diagnosis of mental retardation (including borderline or mild mental retardation)
* Diagnosis of autism, Asperger's syndrome, or another childhood disorder involving learning or relating to other people
* History of a neurological disorder, including epilepsy, traumatic brain injury with loss of consciousness, coma, stroke, Parkinson's disease, etc.
* Diagnosis of active substance abuse (history of a substance abuse disorder without a current substance abuse problem will not be a criterion for exclusion)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Observational ratings of in-group attentiveness | Measured two times per week for 16 weeks
Observational ratings of in-group attentiveness in non-study groups | Measured at Month 6 follow-up
Changes in knowledge of information about social skills taught in the study | Measured at pre- and post-treatment and at Month 6 follow-up
Changes in ability to demonstrate behavioral skills taught in the study | Measured at pre- and post-treatment and at Month 6 follow-up
Level of social functioning | Measured at pre- and post-treatment and at Month 6 follow-up

SECONDARY OUTCOMES:
Self-efficacy | Measured at pre- and post-treatment and at Month 6 follow-up
Working alliance | Measured at pre- and post-treatment and at Month 6 follow-up
Satisfaction with treatment | Measured at pre- and post-treatment and at Month 6 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Silverstein, PhD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (2):
- United States (2):
  - University Behavioral HealthCare, Monmouth Junction, New Jersey
  - University Behavioral HealthCare, New Brunswick, New Jersey

REFERENCES:
- [Background] Silverstein SM, Hatashita-Wong M, Solak BA, Uhlhaas P, Landa Y, Wilkniss SM, Goicochea C, Carpiniello K, Schenkel LS, Savitz A, Smith TE. Effectiveness of a two-phase cognitive rehabilitation intervention for severely impaired schizophrenia patients. Psychol Med. 2005 Jun;35(6):829-37. doi: 10.1017/s0033291704003356. PMID 15997603
- [Background] Silverstein SM, Spaulding WD, Menditto AA, Savitz A, Liberman RP, Berten S, Starobin H. Attention shaping: a reward-based learning method to enhance skills training outcomes in schizophrenia. Schizophr Bull. 2009 Jan;35(1):222-32. doi: 10.1093/schbul/sbm150. Epub 2008 Jan 22. PMID 18212327